CLINICAL TRIAL: NCT02814071
Title: Early Feeding in Acute Pancreatitis in Children - A Randomised Controlled Trial
Brief Title: Early Feeding in Acute Pancreatitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, oledder, Dr. Oren Ledder, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Early Feeding Pancreatitis
Record Dates: First submitted 2016-05-23; First posted 2016-06-27 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Acute Pancreatitis
Keywords: Early Feeding; Acute Pancreatitis; Pediatric
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting with intravenous fluids (No Intervention): The child will be kept fasted. Intravenous fluids will be at a rate and type as directed by the treating clinician. A low fat oral diet will be commenced once abdominal pain resolves and serum amylase/lipase levels decrease from the peak levels as per treating clinician. In the event that the patient is unable to tolerate oral feeding, tube feeding or parenteral nutrition may be commenced based on the clinical decision of the treating clinician(s). This will be recorded as an adverse event. Patients will be re-trialed on oral feeds once initial limiting symptoms or factors have improved or settled as per treating clinician's discretion
- Early enteral feeding (Experimental): Patients will commence on an unrestricted oral diet within 24 hours of presentation, meeting 50% of EER with a regular diet and no fat restriction for the first 24 hours of enteral feeding. A 75-100% EER is targeted ≥ 24 hours of enteral feeding.If the targeted EER is not met orally, a nasogastric tube will be inserted to provide bolus feeds of a standard formula with standard fat content. If the patient fails to tolerate both oral and bolus nasogastric tube feeding, continuous nasogastric tube feeding will be provided. If all fails, enteral nutrition by nasojejunal tube feeding or parenteral nutrition may be commenced based on the clinical decision. Patients will be re-trialed on oral feeds once initial limiting symptoms or factors have improved or settled.
  Interventions: Other: Early enteral feeding

INTERVENTIONS:
Other: Early enteral feeding — Early enteral feeding as per description
  Arms: Early enteral feeding

SUMMARY:
Acute pancreatitis (AP) in children has an increasing incidence and is at times associated with significant morbidity and mortality. Despite this, there is no high-quality evidence-based treatment for childhood AP and current practice is based entirely on historical approach and extrapolation from adult studies.

In this study, we evaluate the use of early enteral feeding in children with AP. The traditional approach to treating AP relies on fasting and intravenous fluids (or occasionally parenteral nutrition) assuming that this minimizes stimulation of an already inflamed pancreas. Contrary to this, evidence exists that early feeding of patients with AP may be beneficial. Randomized controlled trials of fasting vs. early oral diet in adult patients with mild AP, showed no differences in pain, serum amylase and CRP levels, but also shorter hospital stay in those fed earlier. Further data in adults with severe AP demonstrated that early enteral nutrition was associated with decreased mortality, infections and multiorgan failure. These benefits were lost if enteral nutrition was commenced 48 hour after admission. Suggested explanations for these findings include the possibility that enteral nutrition may maintain integrity and function of intestinal mucosa and reduce gut-origin sepsis.

Historically, nasojejunal (NJ) feeds were felt to be safer than oral or nasogastric feeds in the setting of AP by avoiding cephalic and gastric pancreatic stimulation. NJ feeds require moderately invasive tube insertion under radiographic or endoscopic guidance. Recent data suggest that oral feeding with a low fat diet was as safe as NJ feeding.

Several animal models of AP demonstrate that the exocrine pancreas is resistant to cholecystokinin (CCK) stimulation after the onset of AP, suggesting a mechanism for the lack of concern of exacerbating pancreatitis with enteral feeds.

Considering this data it is less certain that diet and fat restriction contribute to treatment of AP. To further challenge the prior conceptions of AP management it is necessary to explore the use of unrestricted diet (full fat) in mild-moderate pediatric AP, a population with recognized low complication risk.

Despite the mounting evidence to the contrary, it is still standard clinical practice to fast children with AP, and only slowly reintroduce feeds depending on the clinical improvement. This is largely due to the lack of clinical interventional studies in children with AP.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial in children with acute pancreatitis, which aims to demonstrate that, compared with the current standard approach of fasting with intravenous fluids, early enteral (oral or nasogastric) feeding with standard diet or formula will improve the following measures of outcome:

1. Length of hospital admission.
2. Serum amylase, lipase, electrolytes, calcium, magnesium, phosphate, urea, creatinine, liver function tests, C-reactive protein (biomarker of inflammation), and full blood count - routine blood tests performed daily until normalisation of serum lipase or until discharge and as directed by treating clinician thereafter.
3. Weight at presentation and "ready for discharge", and at day 30 post-discharge clinic review.
4. Systemic complications including hemodynamic instability, renal failure, intensive care admission.
5. Analgesic requirement.
6. Local complications including pancreatic necrosis, abscess, pseudocyst.
7. Abdominal ultrasound findings during hospital admission (or other abdominal imaging as directed by treating clinicians).

At day 30-60 post-discharge, a routine ultrasound (to assess for localized complication(s) e.g. pseudocyst) and clinical follow-up will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute pancreatitis according to international consensus criteria (Morinville et al. JPGN 2012), which requires at least 2 of the 3 following criteria:

   * Abdominal pain compatible with acute pancreatitis
   * Serum amylase and/or lipase ≥ 3 times upper limits of normal
   * Imaging findings consistent with acute pancreatitis Each episode of acute recurrent pancreatitis will be accepted if each episode is distinct, at least 4 weeks apart from previous episode with intervening normalisation of serum amylase and lipase.
2. Age 3-18 years.
3. Hemodynamically stable.
4. Ability to consent and participate in the study and follow study procedures.

Exclusion Criteria:

1. Severe pancreatitis associated with organ dysfunction and requiring intensive care admission at presentation.
2. Biliary cause of pancreatitis including gallstone pancreatitis and choledochal cyst
3. Autoimmune pancreatitis.
4. High grade traumatic pancreatitis including partial or complete disruption of the pancreatic duct.
5. Presence of other conditions restricting enteral nutrition.
6. Different treatment approach taken by treating clinician due to medical reasons.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Time to ready for discharge | Time to ready for discharge- measured from onset of admission to time when medically assessed ready for discharge. Assessed between 5-10 days up to 14 days.

SECONDARY OUTCOMES:
Length of hospital stay | Length of hospital stay- measured from onset of admission until time of actual discharge from hospital. Assessed between 5-10 days up to 14 days.
Time to clinical resolution of acute pancreatitis | Time to clinical resolution of acute pancreatitis- time from onset of hospital admission until painfree and absence of nausea with no need for analgesia or other symptomatic therapy. Assessed between 5-10 days up to 14 days.
Time to biochemical resolution of acute pancreatitis | Time to biochemical resolution of acute pancreatitis- time from onset of hospital admission to resolution of lipase and/or amylase below upper limit of normal. Assessed between 5-10 days up to 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Oren Ledder, Dr., Principal Investigator — Department of Gastroenterology and Nutrition, Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Department of Pediatric Gastroenterology, Sydney Children's Hospital, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No